CLINICAL TRIAL: NCT02406508
Title: An International Multi-center Phase 2 Study to Evaluate the Safety and Efficacy of Sequential Melphalan Hydrochloride for Injection for Use With the Hepatic Delivery System Treatment Followed by Sorafenib in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Sequential Melphalan for Use With Hepatic Delivery System Treatment Followed by Sorafenib in Patients With Unresectable HCC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No enrollment in the study
Sponsor: Delcath Systems Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHP-HCC-201
Record Dates: First submitted 2015-03-23; First posted 2015-04-02 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hepatic Delivery System Treatment followed by Sorafenib (Experimental): Percutaneous hepatic perfusion with melphalan hydrochloride for injection using the Hepatic Delivery System.
  Melphalan hydrochloride is administered at a dose of 3mg/kg ideal body weight once every 6 weeks for a maximum of 3 cycles of treatment.
  After the Melphalan/HDS treatment patients will be treated with sorafenib according to the package prescribing information.
  Interventions: Device: Melphalan/HDS; Drug: Sorafenib

INTERVENTIONS:
Device: Melphalan/HDS
  Other Names: Melphalan/Hepatic Delivery System; Percutaneous hepatic perfusion (PHP)
Drug: Sorafenib
  Other Names: Nexavar

SUMMARY:
This is a single arm, open label, multi-center, phase 2 study to evaluate the safety and efficacy of sequential treatment with Melphalan/HDS followed by sorafenib in patients with unresectable hepatocellular carcinoma (HCC) confined to the liver.

DETAILED DESCRIPTION:
This is a single arm, open label, multi-center, phase 2 study to evaluate the safety and efficacy of sequential treatment with Melphalan/HDS followed by sorafenib in patients with unresectable hepatocellular carcinoma (HCC) confined to the liver.

Eligible patients will receive up to 3 Melphalan/HDS treatments. Each treatment cycle consists of 6 weeks with an acceptable delay for another 2 weeks before next planned treatment. The Melphalan/HDS treatment will be terminated in patients with progressive disease (PD), complete response (CR), and > 8 weeks delay of recovery from toxicity after last PHP treatment.

With the exception of patients with PD, all patients will be treated with sorafenib after completing the Melphalan/HDS treatment. Patients with PD will be managed with standard of care off-study by their treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. HCC diagnosed by tissue or imaging study
2. Unresectable HCC without extrahepatic disease based on CT
3. At least one target lesion. In patients with prior loco-regional therapy, the target lesion(s) must be located in area(s) outside previous treatment
4. Child-Pugh Class A in the absence of hepatoencephalopathy or clinically evident ascites
5. Barcelona Clinic Liver Cancer (BCLC) stage B
6. MELD Score < 15
7. Eastern Cooperative Oncology Group Performance Status 0-1
8. No prior systemic therapy for HCC
9. No prior radiation therapy to the liver including Y90-, I131-based loco-regional therapy. Prior loco-regional therapy based on other technology for HCC, if any, must have been completed at least 4 weeks prior to baseline imaging
10. Age ≥ 18 years
11. Signed informed consent

Exclusion Criteria:

1. Metastatic disease outside of liver
2. Greater than 50% tumor burden in the liver by imaging
3. History of orthotopic liver transplantation, clinical symptoms of portal hypertension, Whipple's procedure, hepatic artery anatomy incompatible with perfusion or known unresolved venous shunting
4. Evidence of ascites on imaging study, or the use of diuretics for ascites
5. Clinically significant encephalopathy
6. History of allergies or known hypersensitivity to any components of melphalan or the components of the Melphalan/HDS system
7. Known hypersensitivity to heparin or the presence of heparin-induced thrombocytopenia
8. Received an investigational agent for any indication within 30 days prior to first treatment
9. Not recovered from side effects of prior therapy to ≤ grade 1 (according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 [NCI CTCAE v. 4.03]). Certain side effects that are unlikely to develop into serious or life-threatening events (e.g. alopecia) are allowed at > grade 1
10. Those with New York Heart Association functional classification II, III or IV; active cardiac conditions including unstable coronary syndromes (unstable or severe angina, recent myocardial infarction), worsening or new-onset congestive heart failure, significant arrhythmias and severe valvular disease must be evaluated for risks of undergoing general anesthesia
11. History or evidence of clinically significant pulmonary disease that precludes the use of general anesthesia
12. Uncontrolled diabetes mellitus, hypothyroidism, or hyperthyroidism
13. Active uncontrolled infection, including Hepatitis B, Hepatitis C infection. Patients with anti-HBc positive, or HBsAg but DNA negative are exception(s)
14. History of bleeding disorders
15. Brain lesions with a propensity to bleed
16. Known esophageal varices at risk of bleeding, including medium or large esophageal or gastric varices, or active peptic ulcer
17. Previous malignancy within 3 years prior to enrollment, except for curatively-treated basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, bladder carcinoma in situ or breast cancer in situ
18. Inadequate hematologic function as evidenced by any of the following:

    * Platelets < 125,000/µL
    * Hemoglobin ≤ 10 g/dL, independent of transfusion or growth factor support
    * Neutrophils < 1,500/µL
19. Serum creatinine > 1.5 mg/dL
20. Inadequate liver function as evidenced by any of the following:

    * Total serum bilirubin ≥ 2.0 mg/dL
    * Prothrombin time International Normalized Ratio (INR) > 1.5
    * Aspartate aminotransferase (AST) or alanine transaminase (ALT) > 5 times ULN
    * Serum albumin < 3.0 g/dL
21. Alcohol consumption within 30 days of first study treatment, or refusing to abstain from alcohol for the duration of study treatment
22. For female subjects of childbearing potential (i.e., have had a menstrual period within the past 12 months): a positive serum pregnancy test (β-human chorionic gonadotropin) within 7 days prior to enrollment; or unwilling or unable to undergo hormonal suppression to avoid menstruation during treatment
23. Sexually active females of childbearing potential and sexually active males with partners of reproductive potential: unwilling or unable to use appropriate contraception from screening until at least 30 days after last administration of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events after treatment with Melphalan/HDS. | 2 years
Number of patients with adverse events after treatment with Sorafenib following treatment with Melphalan/HDS. | 2 years
Objective response rate in percentage of Melphalan/HDS treatment | 2 years
Progression free survival in months of patients receiving Melphalan/HDS treatment followed by Sorafenib | 2 years

OTHER OUTCOMES:
AUC of melphalan after Melphalan/HDS treatment | Baseline - prior to infusion. Infusion period - 10 min, 20 min, End of infusion. Washout period - 10 min, 20 min, 30 min. Post-procedure period - 5 min, 10 min, 15 min, 30 min, 1 hour, 2 hours, 3.5 hours, 5 hours.
  Pharmacokinetic study
Quality of life questionnaires | Baseline, Week 6 of each PHP cycle, Day 1 of every Sorafenib cycle, End of treatment, every 12 weeks in follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Callahan, RN, Study Director — Delcath Systems
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Montefiore Medical Center, New York, New York